CLINICAL TRIAL: NCT03307317
Title: Mirror Neuron Network Dysfunction as an Early Biomarker of Neurodevelopmental Disorder
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180001; 18-CH-0001
Record Dates: First submitted 2017-10-07; First posted 2017-10-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Developmental Delay
Keywords: Near Infrared Spectroscopy; EEG; Functional Brain Activity; Neurodevelopment; Natural History
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult pilots: Healthy adults between the ages of 18-65 years
- AR infants: Infants with 12 months of age (+/- 2 weeks) with one of the following: observed developmental delay, sibling of a child with autism, premature birth, small for gestational age.
- TD infants: Healthy infants with 9 months of age (+/- 2 weeks)

SUMMARY:
Background:

People show changes in brain activity when they watch other people do actions. This may be part of early social and communication skills. Researchers want to understand the stages of normal development of motor observation and imitation in people and how it relates to social development in infants and toddlers.

Objective:

To study the nature of brain activity that underlies typical brain functioning in infants, toddlers, and adults.

Eligibility:

Infants ages 8 12 months

Healthy adults ages 18 65

Design:

Adult participants will have one visit. They will:

Answer questions about their family, like its size and ethnicity.

Answer questions about their own behavior and do a simple motor task.

Have EEG/fNIRS. A damp elastic cap with small sensors will be placed on the head. Participants will observe stimuli, either on a video screen or of a live person. The sensors will be connected to a computer. That will record the participant s brain activity while watching pictures on a screen.

Infant participants will have 2 visits.

Their parents will answer questions about their family.

The parents will fill out forms about their child s development. These will be mailed to them before each visit.

Parents will stay with their infant while study staff does an assessment of the child s communication, motor, and thinking skills.

Infants will have EEG/fNIRS.

Infants who are at risk for developmental delays will come back for another visit when they are about 2 years old. This will repeat the infant visits but it will not include EEG/fNIRS.

Some questionnaires and assessments will be videotaped.

DETAILED DESCRIPTION:
Objective: This investigation has two main objectives: 1) combine two child-friendly brain imaging techniques and stochastic modeling to determine the neural basis for the development of imitation and mimicry in human infants and 2) use machine learning to identify brain activation patterns that predict impairment in imitation and mimicry in infants at risk for social communication disorders.

Study Population: This study will focus on two groups of infants. The first group includes 60 typically developing infants, who will complete the imitation and neuroimaging paradigm between the ages of 9-12 months (+/- 2 weeks) and again at 12 months of age

(+/- 2 weeks). The second group includes 60 infants at increased risk for social communication disorders, including those with motor delay, language delay, preterm birth, or a sibling with an autism spectrum disorder. These infants will complete the imitation and neuroimaging paradigm at 12 months of age (+/- 1 month) as well as a follow up evaluation of social communication skills and developmental status at 24 months of age (+/- 1 month).

Design: We propose to conduct longitudinal studies of changes in EEG and fNIRS correlates of mirror neuron network activity in typical development and infants at risk for social communication delay. We will measure both EEG mu suppression and hemodynamic change over the motor cortex during an established infant action/observation paradigm. At all study visits, infants will also complete developmental assessments that measure abilities in cognitive, motor, language, and social domains.

Outcome measures: Both neuroimaging measures and developmental status will serve as outcomes for this study. For the typically developing infants, change in the neuroimaging metrics (i.e., percent mu suppression, percent oxyhemoglobin change) will be used to

characterize development of the mirror neuron system, while the relation between neuroimaging variables, their trajectories, and developmental ability will be used to develop hypotheses about the role of the mirror neuron network in development of social communication skills. For the infants at risk for social communication disorders, the main outcome will be developmental status, with neuroimaging metrics used as predictors.

ELIGIBILITY:
* INCLUSION CRITIERIA:

Healthy adults

* Age of 18-65 at study entry
* Healthy and good condition as determined by medical history and physical examination

Healthy Infants

* 9 months +/- 2 weeks of age at time of consent
* Healthy and good condition as determined by medical history and physical examination
* Age appropriate development as determined by parent report and exam
* Full term at birth
* Normal weight for gestational age

At Risk Infants

* 12 months +/- 2 weeks at the time of consent
* Must have at least one of the following: observed developmental delay; sibling of a child with autism; premature birth; small for gestational age

EXCLUSION CRITERIA:

Healthy Adults

* Uncorrected auditory impairment
* Uncorrected visual impairment
* Head injury with loss of consciousness
* Inability to provide consent
* Subject has a condition, that in the opinion of the investigator, creates an unacceptable risk for participation

Healthy and At-Risk Infants

* A language other than English as the primary language spoken at home
* Having a medical impairment that interferes with study participation such as having a g-tube, shunt or seizure disorder and inability to hold one s head upright
* Having a known visual impairment
* Having a known auditory impairment

Ages: 9 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult pilots and TD infants will be recruited from a community sample. AR infants will be recruited from local early intervention providers and pediatricians, following procedures of ongoing collaborative studies at NIH.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2030-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Developmental level | Visit 2 for AR group
  Diagnostic status and behavioral scales that reflect child development at different levels: gross motor, fine motor, language and visual reception.
Hemodynamic response function and mu suppression | Visit 1 for Adult Pilot, TD and AR infants; visit 2 for TD infants
  The change in neuroimaging metrics (i.e., percent mu suppression, percent oxyhemoglobin change) will be used to characterize the development of the mirror neuron system.

CONTACTS AND LOCATIONS:
Overall Officials: Amir H Gandjbakhche, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thorpe SG, Cannon EN, Fox NA. Spectral and source structural development of mu and alpha rhythms from infancy through adulthood. Clin Neurophysiol. 2016 Jan;127(1):254-269. doi: 10.1016/j.clinph.2015.03.004. Epub 2015 Mar 20. PMID 25910852
- [Background] Vanderwert RE, Fox NA, Ferrari PF. The mirror mechanism and mu rhythm in social development. Neurosci Lett. 2013 Apr 12;540:15-20. doi: 10.1016/j.neulet.2012.10.006. Epub 2012 Oct 11. PMID 23063953
- [Background] Anderson AA, Smith E, Chowdhry FA, Thurm A, Condy E, Swineford L, Manwaring SS, Amyot F, Matthews D, Gandjbakhche AH. Prefrontal Hemodynamics in Toddlers at Rest: A Pilot Study of Developmental Variability. Front Neurosci. 2017 May 30;11:300. doi: 10.3389/fnins.2017.00300. eCollection 2017. PMID 28611578
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-CH-0001.html